CLINICAL TRIAL: NCT01251133
Title: A Phase III Study to Assess Immunogenicity and Safety of 4th LBVH0101 Vaccination Compared With 4th Hiberix™ Vaccination in Healthy Toddlers Who Completed Primary Vaccination in LG-VHCL002 Study
Brief Title: Immunogenicity and Safety Study of 4th LBVH0101 After the Primary Vaccination in LG-VHCL002 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Soomin Oh/CRA, LG Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LG-VHCL004
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Infectious Disease by Haemophilus Influenzae Type b
Keywords: Communicable Diseases; Infection; Influenza; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases
MeSH Terms: conditions — Communicable Diseases; Infections; Influenza, Human; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases | interventions — HibTITER protein, Haemophilus influenzae

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LBVH0101 (Experimental)
  Interventions: Biological: LBVH0101 (Hib vaccine)
- Hiberix (Active Comparator)
  Interventions: Biological: Hiberix™ Vaccine

INTERVENTIONS:
Biological: LBVH0101 (Hib vaccine) — 0.5mL
  Arms: LBVH0101
Biological: Hiberix™ Vaccine — 0.5mL
  Arms: Hiberix

SUMMARY:
This is a multi-center, comparative, two-arm, parallel-group, single-blind, phase III study to assess immunogenicity and safety of 4th LBVH0101 (Haemophilus influenzae type b tetanus toxoid conjugate vaccine) vaccination compared with 4th Hiberix™ vaccination after the same vaccination with primary one in healthy toddlers who completed the primary vaccination with LBVH0101 or Hiberix™ in LG-VHCL002 study.

DETAILED DESCRIPTION:
Primary objective: This study was purposed to compare and assess immunogenicity of 4th LBVH0101 or Hiberix™ vaccination in toddlers who completed the primary vaccination with LBVH0101 or Hiberix™, respectively, in LG-VHCL002 study.

Secondary objective: This study was purposed to compare and assess safety of 4th LBVH0101 or Hiberix™ vaccination in toddlers who completed primary vaccination with LBVH0101 or Hiberix™ in LG-VHCL002 study. It was also purposed to assess persistence of immunogenicity prior to 4th vaccination in toddlers who completed the primary vaccination with LBVH0101 or Hiberix™, respectively, in LG-VHCL002 study.

ELIGIBILITY:
Inclusion Criteria:

* Were vaccinated with LBVH0101 or Hiberix™ three times in LG-VHCL002 study
* Healthy male and female infants at the age of 12 to 15 months from birth
* The infants and their parents/legally acceptable representative could comply with all of the scheduled visits in the study
* The parents/legally acceptable representative signed the written consent form.

Exclusion Criteria:

* Subject had been vaccinated with 4th shot of Haemophilus influenzae type b
* Subject is scheduled to be administered with any vaccine other than those specified in the protocol as allowed according to the Standard Immunization Schedule, between the 4th vaccination and Completion Visit
* Subject had suffered from any infectious disease caused by Haemophilus influenzae type b
* Subject has fever of ≥ 37.5°C (axillary temperature) at the day of vaccination
* There is a clear or suspected immune function disorder
* Systemic corticosteroid (prednisolone or equivalent > 0.5 mg/kg/day) was administered for more than 14 days within 30 days prior to administration of the test vaccine or any systemic immunosuppressant was used

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Percentage of the subjects who obtained protective Ab response with anti-PRP Ab titer ≥ 1 ㎍/mL after 4th vaccination | at 4 weeks after 4th vaccination

SECONDARY OUTCOMES:
Percentage of the subjects who maintained preventive Ab response with anti-PRP Ab titer ≥ 1㎍/mL prior to 4th vaccination
Percentage of the subjects who maintained preventive Ab response with anti-PRP Ab titer ≥ 0.15㎍/mL prior to 4th vaccination
Percentage of the subjects who obtained preventive Ab response with anti-PRP Ab titer ≥ 0.15㎍/mL after 4th vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Ansan Hospital, Ansan, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim KH, Kim YK, Kim NH, Chang SH, Lee J, Park EA, Park SE, Eun BW, Lee H, Lee HJ. Immunogenicity and safety of LBVH0101, a new Haemophilus influenzae type b tetanus toxoid conjugate vaccine, compared with Hiberix in Korean infants and children: a randomized trial. Vaccine. 2012 Feb 27;30(10):1886-94. doi: 10.1016/j.vaccine.2011.12.122. Epub 2012 Jan 13. PMID 22245607